CLINICAL TRIAL: NCT06235138
Title: Jawline Improvement Using Patient-specific Angle Implants With Virtual Planning in Orthognathic Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23IUFC01
Record Dates: First submitted 2024-01-11; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-12

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Jawline improvement is nowadays a strong patients' demand. Among patients undergoing orthognathic surgery, it remains sometimes a challenge to manage angle definition due to the classic mandibular osteotomy trait which mostly allows sagittal mandibular movements but can't modify the ramus height. A few types of osteotomies can be used to improve jawline's shape while correcting malocclusion, but they remain technically difficult and often imply the necessity for bone grafting and/or the use of a specific saw and screwdriver. The advent of computer-assisted surgical planning and computer-aided design/ computer-aided manufacturing (CAD-CAM) techniques for patient-specific implant (PSI) fabrication has enabled new methods for managing the jawline in orthognathic surgery. The aim of this study was to assess jawline improvement with patient-specific angle implants in patients undergoing orthognathic surgery with standard osteotomies.Methods: A virtual simulation of a Le Fort I osteotomy (if needed), a sagittal split ramus osteotomy with patient-specific titanium angle implants, and a genioplasty (if needed) was conducted on a preoperative three-dimensional (3D) model of each patient's skull using ProPlan CMF software (Materialise, Leuven, Belgium). Computer-assisted osteotomy saw-and-drill guides and patient-specific implants (PSIs, titanium plates and angle implants) were produced and used during the surgery. The investigators chose to focus on jawline improvement by comparing the preoperative and the post-operative 3D-photographs using the VECTRA H2 3D imagine system (Canfield Scientific, **).

ELIGIBILITY:
* Inclusion Criteria: patients undergoing orthognathic surgery and jawline correction with patient-specific angle implants at Head and Neck Institute, Nice, France
* Exclusion Criteria: None

Ages: 18 Years to 43 Years | Sex: All
Age Groups: Adult
Study Population: Patients undergoing orthognathic surgery and jawline correction with patient-specific angle implants at Head and Neck Institute, Nice, France
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
The primary outcome of interest was the postoperative aspect and position of the gonial angle | postoperative week 4
  The primary outcome of interest was the postoperative aspect and position of the gonial angle, assessed by 3D-stereophotogrametry
Secondary outcome of interest is patients satisfaction | From post operative week 1 to one year follow-up
  Scale title = échelle de Likert. Maximum score 5 (= not satisfied) / minimum score 1 (= total satisfaction)
Secondary outcome of interest is number and type of complications | From post operative week 1 to one year follow-up
  Secondary outcome of interest is number and type of complications

CONTACTS AND LOCATIONS:
Overall Officials: Olina RIOS, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (2):
- France (2):
  - CHU de Nice, Nice, Alpes Maritimes
  - CHU NICE, Nice, Alpes Maritimes